CLINICAL TRIAL: NCT05263115
Title: An Individualized Stair Climbing Program Versus Traditional Resistance Exercise: Effects on Strength, Power, Functional Performance and Cognition in Older Adults
Brief Title: Stair Climbing Exercise Versus Traditional Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Evelien Van Roie, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S66174
Record Dates: First submitted 2022-02-11; First posted 2022-03-02 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Exercise Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise (Active Comparator): 12-week progressive power-oriented resistance exercise program on leg press machine
  Interventions: Other: Resistance Exercise intervention
- Functional stair and stepping-based exercise (Experimental): 12-week progressive functional weight-bearing stair and stepping-based exercise program
  Interventions: Other: Functional stair climbing and stepping-based exercise intervention

INTERVENTIONS:
Other: Resistance Exercise intervention — 12-week progressive resistance exercise intervention
  Arms: Resistance exercise
Other: Functional stair climbing and stepping-based exercise intervention — 12-week progressive stair climbing and stepping-based exercise intervention
  Arms: Functional stair and stepping-based exercise

SUMMARY:
Current evidence suggests resistance exercise as the primary therapeutic strategy to prevent age-related functional decline. The National Strength and Conditioning Association recently stated that a properly designed resistance exercise program should include power exercises performed at higher velocities in concentric movements with moderate intensities. We should be aware that not all older adults are easily motivated to train in unfamiliar gym-based settings with high subscription fees. Therefore, implementation of traditional gym-based resistance exercise at a large scale has been found to be difficult. Interestingly, we have previously shown that the use of high external loads, which implies the need for specific facility memberships, is not necessary to induce neuromuscular gains. This provides strong support for home-based training intervention strategies. Stair climbing or stepping-based exercise constitute a promising avenue to ameliorate the cost-effectiveness and implementation potential of resistance exercise in older adults. Such exercises can induce muscular activation levels similar to high-load resistance exercise and result in similar or even better gains in muscle mass, strength and power compared to slow-speed resistance exercise when properly designed. However, the (neuro)-muscular effects of stair climbing exercise have never been compared to the more optimal power-oriented resistance exercise, which is the primary aim of this study. The secondary aim of this study is to examine if stair climbing exercise also has beneficial effects on cognition.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Unstable cardiovascular disease
* Neurological disorders
* Cognitive malfunctioning (MoCA < 24)
* Low level of physical function (SPPB < 7)
* Acute infections/fever
* Severe musculoskeletal problems
* Systematic engagement in (resistance) exercise in the 12 months prior to participation

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
F-V profile | Change from baseline in F-v profile at 12 weeks
  Force-velocity profiling is carried out unilaterally (dominant leg) on the pneumatic leg press device (Leg Press CC, HUR, Kokkola, Finland). The test protocol consists of a maximal isometric test (knee joint angle = 85°, hip angle = 55°; 3 attempts of 3s), followed by explosive concentric leg extensions at gradually increasing loads (unloaded, 15%, 30%, 45%, 60%, 75% of the maximal isometric force, 2-3 attempts per load, and additional single repetitions until one-repetition maximum is reached). Mean velocity of the best trial per load is used to estimate the individual F-v relationship through a linear equation. This F-v relationship will be used to examine the exercise-induced adaptations. F0 (maximal force), v0 (maximal velocity), a (the equation's slope), Pmax (maximal power) and the corresponding v and F at Pmax are used for the analyses.

SECONDARY OUTCOMES:
Gait speed | Change from baseline in gait speed at 12 weeks
  The average speed to walk 10m as fast as possible (in m/s)
5-repetition sit-to-stand time | Change from baseline in sit-to-stand performance at 12 weeks
  The time (s) needed to perform 5 sit-to-stand transitions.
5-repetition sit-to-stand power | Change from baseline in sit-to-stand performance at 12 weeks
  The power (watt) needed to perform 5 sit-to-stand transitions.
Stair ascent time | Change from baseline in stair climbing performance at 12 weeks.
  The time (s) needed to ascend a flight of stairs.
Stair ascent power | Change from baseline in stair climbing performance at 12 weeks.
  The power (watt) needed to ascend a flight of stairs.
Countermovement jump height | Change from baseline in countermovement jump height at 12 weeks.
  Jump height (cm) in a countermovement jump
MoCA test score | Change from baseline in Montrial Cognitive Assessment test score at 12 weeks.
  Total score (min 0, max 30, higher scores indicate better performance) on the Montreal Cognitive Assessment test
Digit Span Test score | Change from baseline in Digit Span Test score at 12 weeks.
  Total score (min 0, max 30, higher scores indicate better performance) on the Digit Span Test
Trail Making Test Time | Change from baseline in Trail Making Test at 12 weeks.
  Total duration (s) needed to complete the Trail Making Test.
Stroop Test number of words | Change from baseline in Stroop Test at 12 weeks.
  Total number of words red in 45s in the stroop test.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Movement Sciences, Leuven, Belgium

REFERENCES:
- [Derived] Van Roie E, van Uffelen J, Delecluse C. Stair-Climbing Versus Machine-Based Resistance Exercise to Improve Muscle Power Among Older Adults: A Noninferiority Trial. J Strength Cond Res. 2025 Mar 1;39(3):e496-e505. doi: 10.1519/JSC.0000000000005005. Epub 2024 Nov 26. PMID 39590559